CLINICAL TRIAL: NCT06693648
Title: A Randomized, Double-Blind, Multi-Center, Placebo-Controlled, Trial to Evaluate the Efficacy and Safety of Once Daily Diclofenac Gel AMZ001 in the Treatment of Pain and Symptoms of Knee Osteoarthritis
Brief Title: A Study to Evaluate Efficacy and Safety of AMZ001 for the Treatment of Knee Osteoarthritis Symptoms
Acronym: AMZ001
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Amzell (Industry)
Collaborators: NBCD A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AMZ001-007; 2024-517404-11 (EudraCT Number)
Record Dates: First submitted 2024-11-14; First posted 2024-11-18 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Osteoarthritis of Knee; Osteoarthritis, Knee
Keywords: AMZ001; Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- AMZ001 diclofenac gel (Experimental)
  Interventions: Drug: AMZ001 Diclofenac gel
- Placebo gel (Placebo Comparator)
  Interventions: Drug: Placebo gel

INTERVENTIONS:
Drug: AMZ001 Diclofenac gel — Diclofenac gel applied once daily
  Arms: AMZ001 diclofenac gel
Drug: Placebo gel — Matching placebo gel applied once daily
  Arms: Placebo gel

SUMMARY:
This is a multicenter, randomized, double-blind, placebo-controlled, parallel group, 6-week trial of a formulation of AMZ001 once daily versus placebo once daily.

DETAILED DESCRIPTION:
This is a multicenter, randomized, double-blind, placebo-controlled, parallel group, 6-week trial of a formulation of AMZ001 once daily versus placebo once daily. Participants will be evaluated for osteoarthritis by X-ray images of the knees and one knee will be selected for treatment as the target knee. The study gel will be applied directly to that knee throughout the 6 weeks of the study.

ELIGIBILITY:
Inclusion Criteria:

* Participant is able to read and understand the language and content of the study material, understand the requirements for study visits, and is willing to provide information at the scheduled evaluations and appropriate written informed consent has been obtained.
* Femorotibial osteoarthritis (OA) of the knee, according to the American College of Rheumatology (ACR) clinical and radiographic criteria (Altman et al. 1986)
* Radiological OA grade 2, or 3 of the target knee, using the Kellgren-Lawrence method (Kellgren & Lawrence 1957) as graded by central, independent reading of X-ray obtained during screening, or on a recent (within 6 months) X-ray image which fulfils the specifications for central reading.
* Pain score rated on an 11-point numerical rating scale of the target knee of ≥20 and ≤45 out of 50 in response to the WOMAC pain sub-score (5 questions), at the time of screening and baseline.
* The WOMAC pain sub-score on the target knee must exceed the one on the contralateral knee, regardless of the eligibility of the contralateral knee.
* At screening Visit 1a, participants report that their typical OA knee pain in one or both knees when not using medication is ≥4 out of 10.
* Daily OA knee pain diary average numerical rating scale (NRS) score of ≥4 and ≤9 in the target knee, for the 7 days immediately preceding baseline (Day 1). The average calculation is based on the recorded scores during this entire period with a requirement of at least 4 days of data recorded.
* Women of child-bearing potential must use at least an acceptably effective method of contraception (progestogen-only oral hormonal contraception, where inhibition of ovulation is not the primary mode of action, male or female condom with or without spermicide, cap, diaphragm or sponge with spermicide) from enrolment up to at least 3 months after the study end. Postmenopausal status is defined as being amenorrheic for at least 1 year prior to screening. Sexually active men with a female partner of childbearing potential must agree to use condom from enrolment up to at least 3 months after the study end.
* Knee pain in the target knee for at least 14 days of the preceding month (periarticular knee pain due to OA and not due to non-OA conditions such as bursitis, tendonitis, etc.) based on participant report.
* Except for OA, the participant is in reasonably good health as determined by the Investigator.

Exclusion Criteria:

* Known or suspected hypersensitivity to or previous hypersensitivity reactions to diclofenac or of the excipients in either of the investigational products.
* Patients in whom asthma, angioedema, urticaria, or acute rhinitis are precipitated by acetylsalicylic acid or other non-steroidal anti-inflammatory drugs (NSAIDs).
* Any physical impediment to gel application on the target knee.
* Intra-articular delivery of corticosteroids or hyaluronic acid in the target knee within 6 months of screening or into any other joint within 30 days of screening.
* High dose (equivalent to > 10 mg of prednisone/day) systemic corticosteroid treatment of more than 14 days during the past 6 months prior to screening.
* Major surgery/ arthroscopy of the target knee within the previous year prior to screening or aspiration of effusion of the target knee within 12 weeks prior to enrollment.
* Planned surgery of the target knee within the next 12 months.
* Use of a currently unapproved investigational drug, device or biologic within 3 months prior to screening.
* Presence of concomitant non-osteoarthritic disease affecting either knee, such as rheumatoid arthritis, psoriasis, gout or clinically relevant pseudogout, if there is reason to believe that the disease(s) may significantly interfere with the interpretation of the clinical response to the study drug.
* Perioperative period in the setting of coronary artery bypass graft surgery.
* Current malignancy or treatment for malignancy within the past five years, with the exception of non-melanoma skin cancer, unless affecting the target knee area, or carcinoma in situ events.
* Any other abnormal laboratory results or significant medical conditions that the Investigator believes should preclude the participant's participation in the trial.
* Secondary OA of the target knee, previous procedures or trauma affecting joint homeostasis including total meniscectomy or septic arthritis, or any other serious condition leading to secondary OA of the target knee.
* Reported incidence of any of the following diseases: known OA of the hip(s) if pain in either or both hip(s) exceeds that of the target knee using the WOMAC hip pain subscore, or presence of significant radicular back pain.
* Presence of severe pain in either knee, defined as > 45 out of 50 in response to the WOMAC pain sub-score (5 questions), at the time of screening and baseline, regardless of the eligibility of the contralateral knee.
* Presence of a defined cut-off of pain variability during the screening period of 1.5 out of 10:
* Pain Numeric Rating Scale (NRS) scores must be recorded for the target knee on at least 4 out of the 7 days immediately preceding baseline (Day 1)
* Observed standard deviation of the Daily osteoarthritis (OA) knee pain diary average NRS intensity score for 7 days immediately preceding baseline (Day

  1) must not exceed 1.5
* Body mass index > 45.0 kg/m2.
* Estimated glomerular filtration (eGFR) rate < 30 mL/min using the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI 2021) formula.
* Generalized skin irritation, previous skin reactions upon use of topical NSAIDs, current skin irritation or redness at the planned site of gel application, or significant skin disease including psoriasis, as judged by the investigator.
* Use of any topical medication on the planned application site within 15 days of the time of randomization.
* Use of moderate or higher strength of opioid medication for the treatment of pain within 6 weeks before the screening visit.
* Use of duloxetine, pregabalin, or gabapentin within 4 weeks before the screening visit.
* History of alcohol or drug abuse within the past year prior to randomization.
* Pregnant and breastfeeding women are excluded for participation.

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 540 (Estimated)
Dates: Start 2025-02-18 (Actual); Primary Completion 2025-12-22 (Actual); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in the WOMAC pain sub-score in the target knee at week 2. | Baseline and Week 2
  WOMAC: Western Ontario and McMasters University Osteoarthritis Index Scale: 0-100, 100 being the worse

SECONDARY OUTCOMES:
Change from baseline in the WOMAC pain sub-score at week 1, in the target knee | Baseline and Week 1
  WOMAC: Western Ontario and McMasters University Osteoarthritis Index Scale: 0-100, 100 being the worse
Change from baseline in daily pain at Day 8 using an 11-point Numeric Rating Scale (NRS) | Baseline and Day 8
  NRS: Numeric Rating Scale Scale: 0 -10, 10 being the worse
Change from baseline in daily pain at Day 7 using an 11-point Numeric Rating Scale (NRS) | Baseline and Day 7
Change from baseline in daily pain at Day 6 using an 11-point Numeric Rating Scale (NRS) | Baseline and Day 6
Change from baseline in daily pain at Day 5 using an 11-point Numeric Rating Scale (NRS) | Baseline and Day 5
Change from baseline in daily pain at Day 4 using an 11-point Numeric Rating Scale (NRS) | Baseline and Day 4
Change from baseline in daily pain at Day 3 using an 11-point Numeric Rating Scale (NRS) | Baseline and Day 3
Change from baseline in daily pain at Day 2 using an 11-point Numeric Rating Scale (NRS) | Baseline and Day 2
Change from baseline in daily pain at Day 1 using an 11-point Numeric Rating Scale (NRS) | Baseline and Day 1

CONTACTS AND LOCATIONS:
Locations (11):
- United States (7):
  - Millennium Clinical Trials, Thousand Oaks, California
  - Eastern Research Inc, Hialeah, Florida
  - Future Medical Research, Longwood, Florida
  - DelRicht Research, New Orleans, Louisiana
  - DelRicht Research, Rockville, Maryland
  - Oakland Medical Research, Troy, Michigan
  - West Clinical Research, Morehead City, North Carolina
- hong Kong Center for Clinical Research, Hong Kong, China
- Charles University, Prague, Czechia
- Sanos Clinic, Herlev, Denmark
- Medyczne Centrum Hetmanska Piotr Leszczynski, Poznan, Poland

IPD SHARING:
Plan to Share IPD: Undecided